CLINICAL TRIAL: NCT05103163
Title: The Effect of Foot Reflexology on Patient Satisfaction, Pain, and Vital Signs After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gurkan Kapikiran (Other)
Responsible Party: Sponsor-Investigator, Gurkan Kapikiran, Assistant Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/2
Record Dates: First submitted 2021-10-03; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Surgery
Keywords: Abdominal Surgery; Foot Reflexology; Vital Signs; Patient Satisfaction; Pain
MeSH Terms: conditions — Patient Satisfaction; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Which of the patients included in the study would be in the experimental group and which would be in the control group was determined according to the randomization table determined by the web-based random assignment software (RAY). There are two columns in the table as group 1 and group 2. Which column would be in the experimental group and which would be in the control group was determined by drawing lots. As a result of the draw, it was determined that group 1 would be in the control group and group 2 would be in the experimental group. Then, group assignments were made in accordance with the randomization order determined by RAY.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot reflexology group (Experimental): Before the reflexology application, a personal information form was applied to the patients who had abdominal surgery. As a pre-test, satisfaction levels in terms of pain and nursing were evaluated. Then, vital signs (systolic blood pressure, diastolic blood pressure, pulse, respiration and saturation) were measured. Foot warming movements were started and then the warming movements were terminated by applying pressure to the solar plexus area of the left foot. Then in order; Reflexology was applied to the brain, lymphatic system, blood pressure area, lung, adrenal gland, thyroid, diaphragm, stomach and joint areas. Afterwards, relaxation movements were made for the foot, pressure was applied to the solar plexus and the reflexology application was completed within 30 minutes. Immediately after the application, vital signs were re-measured as a post-test, and the numerical pain scale and care satisfaction scale were applied again.
  Interventions: Other: Foot Reflexology
- No treatment group (No Intervention): To the patients in the control group; Personal Information Form, Numerical Pain Scale (NPS) and Newcastle Nursing Care Satisfaction Scale (NNCSS) were applied as pre-test. After the questions were answered, NNCSS with NPS was applied again 40 minutes later as a final test, without any intervention other than the clinical protocol.

INTERVENTIONS:
Other: Foot Reflexology — Reflexology application is an energy balancing system with its own pressure technique that provides recovery by rubbing the reflex (nerve endings) points, stroking and applying pressure during squeezing movements. Thanks to the pressure and massage applie
  Arms: Foot reflexology group

SUMMARY:
Reflexology practice is an effective method in pain control by stimulating the release of endorphins. The study was conducted to determine the effect of foot reflexology applied to patients undergoing abdominal surgery on pain, patient satisfaction and vital signs. The study was conducted in a randomized controlled manner. The population of the study consisted of adult patients who underwent abdominal surgery in a university hospital in Turkey. The sample consisted of 156 patients with the indicated power analysis, including the analysis 78 experimental and 78 controls. Data were collected between October 2020 and May 2021 using Personal Information Form, Numerical Pain Scale, Newcastle Nursing Care Satisfaction Scale and Vital Signs Registration Form.

DETAILED DESCRIPTION:
This study was conducted in a randomized controlled experimental setup. This research was conducted in the general surgery clinic of a university hospital in Turkey between October 2020 and May 2021.

The universe of the research; consisted of 261 patients aged 18 years and over who underwent abdominal surgery in the general surgery ward of a university hospital. The G Power 3.1.9.7 computer program was used to calculate the sample size. According to this program, it was determined that a total of 156 patients, 78 patients in each group, should be reached, with an effect size of 0.4, a margin of error of 0.04, a confidence interval of 0.95, and a population representation power of 95%. 57 patients who did not meet the inclusion criteria and 48 patients who did not volunteer to participate in the study were not included in the sample.

Which of the patients included in the study would be in the experimental group and which would be in the control group was made according to the randomization table determined by the web-based random assignment software (RAY). There are two columns in the table as group 1 and group 2. Which column would be in the experimental group and which would be in the control group was determined by drawing lots. As a result of the draw, it was determined that group 1 would be in the control group and group 2 would be in the experimental group. Then, group assignments were made in accordance with the randomization order determined by RAY.

In the collection of data; "personal information form", "numerical pain scale", "newcastle nursing care satisfaction scale" and vital signs registration form were used.

Data were collected by the first researcher by face-to-face interview method between October 2020 and May 2021. Patients who met the inclusion criteria were recruited three days a week and on weekends after surgery.

A single post-operative session (30 minutes) of foot reflexology was applied to patients with abdominal surgery in the intervention group by the first investigator who had received reflexology practice training before starting the study. Patient privacy was respected in all procedures. During the application, it was ensured that the ambient sounds were as quiet and calm as possible. The monitor and phones were set to silent mode, and the television was turned off during the application. The bed-ends were removed, the patient was asked to lie in the supine position, and the investigator supported the patient's feet with a pillow, ready for reflexology. After these preparations, the researcher washed and dried his hands, took some olive oil, rubbed his hands and brought it to body temperature. Personal information form was applied before the reflexology application. As a pre-test, pain and nursing satisfaction levels were evaluated with newcastle nursing care satisfaction scale. Then, vital signs (systolic blood pressure, diastolic blood pressure, pulse, respiration and saturation) were measured. Foot warming movements, which is the first stage of foot reflexology, were applied to the left foot for 5 minutes. As foot warming movements; Achilles tendon stretching, rotation, executing the thumbs of the hand under the foot, bilateral wrist loosening and laundry tightening were performed using several methods. Then, the warm-up movements were terminated by applying deep and painless pressure to the solar plexus area of the left foot for 1 minute. Then in order; Reflexology was applied to the brain (pineal and pituitary region in the thumb, hypothalamus), lymphatic system, tension region (projection of the solar plexus on the foot), lung, adrenal gland, thyroid, diaphragm, stomach and joint regions. Afterwards, relaxation movements were made for the foot, pressure was applied to the solar plexus and the reflexology application was completed within 30 minutes. Immediately after the application, vital signs were re-measured as a post-test, and numerical pain scale and newcastle nursing care satisfaction scale were re-applied.

To the patients in the control group; personal information form, numerical pain scale and newcastle nursing care satisfaction scale were used as pre-tests. After the questions were answered, numerical pain scale and newcastle nursing care satisfaction scale were re-administered 30 minutes later as a post-test without any intervention other than the clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above who are open to communication,
* Hospitalized for at least two nights
* Defining the severity of pain as 4 and above,
* Any lesion, wound, infection, etc. that prevents the practice of standing reflexology. non,
* Not diagnosed with cancer
* Deep vein thrombosis, epilepsy, Thrombophlebitis, febrile diseases etc. without diseases,

Exclusion Criteria:

* Presence of any lesion, wound, infection etc. on the foot
* Presence of deep vein thrombosis
* Presence of epilepsy
* With thrombophlebitis and febrile diseases
* Those who do not volunteer to participate in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 0-30 minutes
  It is a Likert-type scale, scored between 1 and 5, consisting of 19 questions containing patients' views of satisfaction with nursing care.
Pain Level | 0.-30. minutes
  It is a numeric scale which is based on explaining pain severity with numbers, and where 0 point means no pain and 10 points mean unbearable pain
Blood pressure measurement | 0.-30. minutes
  Systolic blood pressure was measured with a digital sphygmomanometer (mm Hg).
Blood pressure measurement | 0.-30. minutes
  Diastolic blood pressure was measured with a digital sphygmomanometer (mm Hg).
Pulse measurement | 0.-30. minutes
  The patient's heart rate in 1 minute was measured.
Respiratory rate measurement | 0.-30. minutes
  The respiratory rate of the patient in 1 minute was measured.
oxygen saturation measurement | 0.-30. minutes
  Oxygen saturation was measured with a pulse oximeter device.

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided